CLINICAL TRIAL: NCT06192017
Title: Development of a Molecular Diagnostic Tool for Endometrial Cancer.
Status: Completed | Type: Observational
Sponsor: MiMARK Diagnostics, S.L. (Industry)
Collaborators: Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Other Study IDs: WomEC SEGO
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Endometrium Cancer
Keywords: Endometrial Cancer, EC
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Uterine Aspirate Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Post-menopausal women with AUB: The patients will be divided into different study groups: "Control" and cases or "EC", the latter could be subdivided and analyzed in separate groups related to their prognosis. The "Control" patients are those patients with symptoms compatible with endometrial cancer but who are diagnosed with benign and / or healthy pathology; while "EC" patients present associated symptoms and are diagnosed with endometrial cancer.
  Interventions: Diagnostic Test: WomEC

INTERVENTIONS:
Diagnostic Test: WomEC — The study will collect pipelle biopsies from post-menopausal women presenting with AUB entering to the EC diagnostic process at the clinical consultancy or emergency room. In the study an endometrial biopsy by aspiration will be collected (i.e., pipelle biopsy) and it will be used for (1) diagnostic purposes following current procedures (i.e., pathological examination and diagnosis); (2) placed in a collection tube for WomEC test.

SUMMARY:
WomEC is an in vitro diagnostic test for Endometrial Cancer (EC) based on the detection of the expression level of a combination of 5 proteins in the soluble fraction of a pipelle biopsy specimen. The aim of the study consists in validating WomEC's ELISA test, creating and freezing an algorithm to rule out EC in post-menopausal women with abnormal uterine bleeding (AUB).

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (≥1 year without menstruation) with AUB who present with:

  1. Endometrium > 3mm by transvaginal ultrasound, OR
  2. Endometrium ≤ 3mm who meet at least one of the following criteria:

  i. Persistent symptoms (more than one episode of metrorrhagia) ii. Heterogenous endometrium on transvaginal ultrasonography iii. Risk factors (BMI ≥ 30, use of tamoxifen, hormone replacement therapy (HRT), Lynch syndrome, BRCA mutation.
* Obtaining written informed consent

Exclusion Criteria:

* Women with an active pelvic infection.
* Women who have had viral infections with evidence of active and latent disease such as Hepatitis B, Hepatitis C, and HIV infection. Patients who have had Hepatitis C in the past but who have been successfully treated and in whom viral replication has not been observed in the last year will be included.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — (Adult, Older Adult)
Study Population: Post-menopausal women presenting AUB entering to the EC diagnostic process at the clinical consultancy or emergency room.
Sampling Method: Probability Sample
Enrollment: 1950 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Regulatory Requirements Study | 12 months
  Ensure the stability of the samples under defined conditions (pre-analytica) and the analytical validation of the developed WomEC's ELISA test.
Algorithm training with Proprietary Antibodies | 12 months
  Train the current WomEC's algorithms defined in MS by assessing the clinical performance of different EC biomarkers individually and in combination to rule out EC in post- menopausal women with AUB using MiMARK's proprietary antibodies.
Algorithm testing and freeze | 12 months
  To test and freeze the defined algorithm measured with MiMARK's antibodies to rule out EC in post-menopausal women with AUB.

SECONDARY OUTCOMES:
To determine the accuracy of WomEC alone for the diagnosis of EC by pipelle biopsy. | 12 months
  Test the ability of WomEC to discriminate between EC and non-EC patients.
Evaluation of the performance of different models of WomEC to determine histological subtype. | 12 months
  Calculate the sensitivity, specificity, accuracy, precision, and clinical validity of WomEC to determine an histological subtype.
Evaluation of the performance of WomEC to determine other prognostic factors of EC. | 12 months
  Calculate the sensitivity, specificity, accuracy, precision, and clinical validity of WomEC to determine other prognostic factors of EC.
Evaluation of the performance of WomEC to diagnose endometrial atypical hyperplasia. | 12 months
  Calculate the sensitivity, specificity, accuracy, precision, and clinical validity of WomEC to diagnose endometrial atypical hyperplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil-Moreno, MD, PhD, Principal Investigator — Hospital Universitari Campus Vall d'Hebron
Locations (26):
- Spain (26):
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Dexeus - Quirón de Barcelona, Barcelona, Barcelona
  - Hospital Universitari Campus Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Universitario de Igualada, Igualada, Barcelona
  - Hospital Universitari de Bellvitge - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de la Plana, Villarreal, Castellon
  - Hospital Clínico de Santiago, A Coruña, Galicia
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital General Universitari de València, Valencia, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia, Valencia
  - Hospital Universitario de Puerto Real, Cadiz
  - Hospital General Universitari de Castelló, Castellon
  - Hospital Universitario de León, León
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Dueholm M, Hjorth IMD, Dahl K, Hansen ES, Ortoft G. Ultrasound Scoring of Endometrial Pattern for Fast-track Identification or Exclusion of Endometrial Cancer in Women with Postmenopausal Bleeding. J Minim Invasive Gynecol. 2019 Mar-Apr;26(3):516-525. doi: 10.1016/j.jmig.2018.06.010. Epub 2018 Jun 23. PMID 29944932
- [Background] Clarke MA, Long BJ, Del Mar Morillo A, Arbyn M, Bakkum-Gamez JN, Wentzensen N. Association of Endometrial Cancer Risk With Postmenopausal Bleeding in Women: A Systematic Review and Meta-analysis. JAMA Intern Med. 2018 Sep 1;178(9):1210-1222. doi: 10.1001/jamainternmed.2018.2820. PMID 30083701
- [Background] van Hanegem N, Prins MM, Bongers MY, Opmeer BC, Sahota DS, Mol BW, Timmermans A. The accuracy of endometrial sampling in women with postmenopausal bleeding: a systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2016 Feb;197:147-55. doi: 10.1016/j.ejogrb.2015.12.008. Epub 2015 Dec 19. PMID 26748390
- [Background] Bradley LD. Complications in hysteroscopy: prevention, treatment and legal risk. Curr Opin Obstet Gynecol. 2002 Aug;14(4):409-15. doi: 10.1097/00001703-200208000-00008. PMID 12151831
- [Background] Helpman L, Kupets R, Covens A, Saad RS, Khalifa MA, Ismiil N, Ghorab Z, Dube V, Nofech-Mozes S. Assessment of endometrial sampling as a predictor of final surgical pathology in endometrial cancer. Br J Cancer. 2014 Feb 4;110(3):609-15. doi: 10.1038/bjc.2013.766. Epub 2013 Dec 24. PMID 24366295
- [Background] Visser NCM, Reijnen C, Massuger LFAG, Nagtegaal ID, Bulten J, Pijnenborg JMA. Accuracy of Endometrial Sampling in Endometrial Carcinoma: A Systematic Review and Meta-analysis. Obstet Gynecol. 2017 Oct;130(4):803-813. doi: 10.1097/AOG.0000000000002261. PMID 28885397
- [Background] Colas E, Perez C, Cabrera S, Pedrola N, Monge M, Castellvi J, Eyzaguirre F, Gregorio J, Ruiz A, Llaurado M, Rigau M, Garcia M, Ertekin T, Montes M, Lopez-Lopez R, Carreras R, Xercavins J, Ortega A, Maes T, Rosell E, Doll A, Abal M, Reventos J, Gil-Moreno A. Molecular markers of endometrial carcinoma detected in uterine aspirates. Int J Cancer. 2011 Nov 15;129(10):2435-44. doi: 10.1002/ijc.25901. Epub 2011 Apr 8. PMID 21207424
- [Background] Perez-Sanchez C, Colas E, Cabrera S, Falcon O, Sanchez-del-Rio A, Garcia E, Fernandez-de-Castillo L, Muruzabal JC, Alvarez E, Fiol G, Gonzalez C, Torrejon R, Moral E, Campos M, Repolles M, Carreras R, Jimenez-Lopez J, Xercavins J, Aibar E, Perdones-Montero A, Lalanne E, Palicio M, Maes T, Rosell-Vives E, Nieto C, Ortega A, Pedrola N, Llaurado M, Rigau M, Doll A, Abal M, Ponce J, Gil-Moreno A, Reventos J. Molecular diagnosis of endometrial cancer from uterine aspirates. Int J Cancer. 2013 Nov 15;133(10):2383-91. doi: 10.1002/ijc.28243. Epub 2013 Jun 21. PMID 23649867
- [Background] Martinez-Garcia E, Lopez-Gil C, Campoy I, Vallve J, Coll E, Cabrera S, Ramon Y Cajal S, Matias-Guiu X, Van Oostrum J, Reventos J, Gil-Moreno A, Colas E. Advances in endometrial cancer protein biomarkers for use in the clinic. Expert Rev Proteomics. 2018 Jan;15(1):81-99. doi: 10.1080/14789450.2018.1410061. Epub 2017 Nov 30. PMID 29183259
- [Background] Martinez-Garcia E, Lesur A, Devis L, Campos A, Cabrera S, van Oostrum J, Matias-Guiu X, Gil-Moreno A, Reventos J, Colas E, Domon B. Development of a sequential workflow based on LC-PRM for the verification of endometrial cancer protein biomarkers in uterine aspirate samples. Oncotarget. 2016 Aug 16;7(33):53102-53115. doi: 10.18632/oncotarget.10632. PMID 27447978
- [Background] Martinez-Garcia E, Lesur A, Devis L, Cabrera S, Matias-Guiu X, Hirschfeld M, Asberger J, van Oostrum J, Casares de Cal MLA, Gomez-Tato A, Reventos J, Domon B, Colas E, Gil-Moreno A. Targeted Proteomics Identifies Proteomic Signatures in Liquid Biopsies of the Endometrium to Diagnose Endometrial Cancer and Assist in the Prediction of the Optimal Surgical Treatment. Clin Cancer Res. 2017 Nov 1;23(21):6458-6467. doi: 10.1158/1078-0432.CCR-17-0474. Epub 2017 Aug 8. PMID 28790116
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- [Background] Fawcett T. An introduction to ROC analysis. Pattern Recognit Lett. North-Holland; 2006;27:861-74.
- [Background] Robin X, Turck N, Hainard A, Tiberti N, Lisacek F, Sanchez JC, Muller M. pROC: an open-source package for R and S+ to analyze and compare ROC curves. BMC Bioinformatics. 2011 Mar 17;12:77. doi: 10.1186/1471-2105-12-77. PMID 21414208